Translating Research Into Practice: A Regional Collaborative to Reduce Disparities in Breast Cancer Care

Information Sheet for Key Informant Interviews NCT03514433

Tracy.Battaglia@bmc.org 11-21-2019.

## BOSTON MEDICAL CENTER AND THE BOSTON UNIVERSITY SCHOOLS OF MEDICINE, PUBLIC HEALTH AND DENTAL MEDICINE





## RESEARCH INFORMATION SHEET FOR KEY INFORMANT INTERVIEWS

You are being asked to voluntarily participate in a research study. We are doing this study to learn more about the experiences of Patient Navigators and other hospital staff across Boston who are all participating in the same city-wide breast cancer navigation program. The purpose is to see what is easy and what is difficult about doing navigation work at each of the participating hospitals. If you agree, we will interview you to learn more about your navigation work and involvement in TRIP, and then ask you to complete a 1-page survey about yourself. It will ask about your race, ethnicity, education background, and current role. You may choose to answer some or all of the questions in the interview and the survey. You will receive \$50 in the form of a reloadable debit card for your participation.

We will make an audio recording of the interviewer's questions and your responses. If you ask us not to, we won't record you. You can skip questions that you do not want to answer, or stop the interview at any time. Your participation in this interview will have no effect on performance reviews.

We will not record your name or other directly identifiable information in the study data, but we may record details about your institution and role. These details could possibly identify you. We will store your information in ways we think are secure. We will store paper files in locked filing cabinets. We will store electronic files in computer systems that are protected by passwords and encryption. However, we cannot promise complete confidentiality.

This study is covered by a Certificate of Confidentiality (CoC) from the National Institutes of Health. All studies funded by the National Institutes of Health that involve identifiable information are covered by a CoC. The CoC provides how we can share research information. Because the study has a CoC, we cannot give out research information that may identify you to anyone that is not involved in the research or overseeing the research except as we describe below. Even if someone tries to get your information in connection with a legal proceeding, we cannot give it to them. The CoC does not prevent you from sharing your own research information or asking us to share your information.

We will share research data where we have removed anything that we think would show your identity. There still may be a small chance that someone could figure out that the information is about you. Such sharing includes:

- Publishing results in a book or journal.
- Adding results to a Federal government database.
- Using research data in future studies, done by us or by other scientists.

If you have any questions, please contact Tracy Battaglia, the lead Principal Investigator at Tracy.Battaglia@bmc.org or (617) 638-8036.